CLINICAL TRIAL: NCT04185545
Title: Efficacy, Safety and Immunogenicity of Rotavirus RV3 Vaccine (Bio Farma) in Neonates, Lot to Lot Consistency and Antigen Interference With Co-Administered EPI Vaccines (Phase III)
Brief Title: Efficacy, Safety and Immunogenicity of Rotavirus RV3 Vaccine (Bio Farma) in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RV 0319
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Rotavirus; Vaccine
MeSH Terms: interventions — RV3 rotavirus vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 1 (Experimental): 3 oral doses of RV3 vaccine (Bio Farma) batch 1; administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Biological: Rotavirus RV3 Vaccine (Bio Farma)
- Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 2 (Experimental): 3 oral doses of RV3 vaccine (Bio Farma) batch 2; administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Biological: Rotavirus RV3 Vaccine (Bio Farma)
- Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 3 (Experimental): 3 oral doses of RV3 vaccine (Bio Farma) batch 3; administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Biological: Rotavirus RV3 Vaccine (Bio Farma)
- Immunogenicity Group - Placebo (Placebo Comparator): 3 oral doses of Placebo; administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Other: Placebo
- Other Efficacy Group - RV3 Vaccine (Bio Farma) (Experimental): 3 oral doses of RV3 vaccine (Bio Farma) administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Biological: Rotavirus RV3 Vaccine (Bio Farma)
- Other Efficacy Group - Placebo (Placebo Comparator): 3 oral doses of Placebo administered at 0-5 days, 8-10 weeks, and 12-14 weeks of age.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Rotavirus RV3 Vaccine (Bio Farma) — Each 1 mL dose of the final product of oral liquid rotavirus vaccine contains > 5x10^6 fcfu/mL rotavirus vaccine strain RV3
  Arms: Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 1; Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 2; Immunogenicity Group - RV3 Vaccine (Bio Farma) Batch 3; Other Efficacy Group - RV3 Vaccine (Bio Farma)
Other: Placebo — Each 1 mL dose of placebo contains 30% of sucrose in DMEM
  Arms: Immunogenicity Group - Placebo; Other Efficacy Group - Placebo

SUMMARY:
This phase III trial aims to assess the efficacy, safety and immunogenicity of Rotavirus RV3 Vaccine (Bio Farma) in neonates, lot-to-lot consistency, and antigen interference with co-administered EPI vaccines

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study to investigate the efficacy, safety and immunogenicity following three doses of rotavirus RV3 vaccine (Bio Farma) administered as a neonatal schedule

ELIGIBILITY:
Inclusion Criteria:

1. Neonate 0-5 days (0-144 hours) of age at the time of first dose.
2. Neonate is in good health as determined by clinical judgment, including a medical history and physical exam, which confirms the absence of a current or past disease state considered significant by the investigator.
3. The neonate was born full term (minimum of 37 completed weeks and maximum of 42 completed weeks gestation).
4. Neonate birth weight 2500-4000 g inclusive.
5. Parent or guardian has been informed properly regarding the study and signed the informed consent form.
6. Parent or guardian commits to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. The subject has direct relatives relationship with the study team.
3. The subject has evolving mild, moderate or severe illness, especially infectious diseases or fever (body temperature 37.5°C) within the 48 hours preceding enrollment.
4. Subject with a known or suspected history of allergy to any component of the vaccines (based on anamnesis).
5. Subject with a biological mother with a known or suspected human immunodeficiency virus (HIV) or Hepatitis B infection.
6. Subject with known or suspected major congenital malformations or genetically determined disease.
7. Subject with intussusception.
8. Subject with a known or suspected disease of uncontrolled coagulopathy or blood disorders contraindicating for phlebotomy.
9. Subject with a known or suspected disease of the immune system or those who have received immunosuppressive therapy, including immunosuppressive courses of systemic corticosteroid.
10. Subject who have ever received any blood products, including immunoglobulin, or for whom receipt of any blood product is anticipated during the course of study.
11. Any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
12. Subject immunized with non-EPI vaccines.
13. Gastroenteritis in the 24 hours preceding dosing (temporary exclusion criteria).
14. Subject planning to move from the study area before the end of the study period.

Ages: 1 Minute to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of three doses against severe acute rotavirus gastroenteritis | 2 weeks after three doses to 18 months of age
  Episodes of severe rotavirus gastroenteritis (defined as a modified Vesikari score ≥ 11 and rotavirus antigen detected in stool by ELISA)

SECONDARY OUTCOMES:
Efficacy of three doses against rotavirus gastroenteritis of any severity and all-cause gastroenteritis | 2 weeks after three doses to 18 months of age
  Episodes of rotavirus gastroenteritis of any severity (based on modified Vesikari score and rotavirus antigen detected in stool by ELISA) and all-cause gastroenteritis
Serum immune response (sIgA) after third dose | 28 days after the third dose
  Percentage of subjects with ≥ 3 times increase in serum anti-rotavirus IgA (sIgA) from baseline to 28 days after the third dose
Stool excretion following each dose | 3-5 days after each dose
  Detectable RV3 excretion in stool (by PCR) any day from day 3 to day 5 following each dose
Cumulative serum immune response | 28 days after each dose
  Cumulative serum anti-rotavirus IgA (sIgA) following each dose
Lot to lot consistency | 28 days after the third dose
  Percentage of subjects with ≥ 3 times increase in serum anti-rotavirus IgA (sIgA) from baseline to 28 days after the third dose
Solicited and unsolicited adverse events (AE) | Up to 28 days after the third dose
  Number of solicited and unsolicited Adverse Events (AE), from randomization to 28 days following last dose
Serious adverse events (SAE) | Up to 28 days after the third dose
  Number of Serious Adverse Events (SAE), from randomization to 28 days following last dose
Serum immune response (sIgA) after the first dose | 28 days after the first dose
  Percentage of subjects with ≥ 3 times increase in serum anti-rotavirus IgA (sIgA) from baseline to 28 days after the first dose
Serum immune response (sIgA) after the second dose | 28 days after the second dose
  Percentage of subjects with ≥ 3 times increase in serum anti-rotavirus IgA (sIgA) from baseline to 28 days after the second dose
Abnormality of ALT and AST levels | 28 days after the first dose
  Abnormality of ALT and AST levels measured 28 days following first dose, assessed as probably or definitely related to the dosing
Immune interference | 28 days after non-EPI vaccination
  Percentage of subjects with reciprocal titre ≥ 1:8 against poliovirus strains 1-3 measured 28 days after bOPV4+ IPV and Pentabio 3 vaccination
Geometric Mean Titre (GMT) | 28 days after each dose
  Geometric Mean Titre (GMT) of serum IgA 28 days after each dose
Serum neutralizing antibodies (SNA) after the third dose | 28 days after the third dose
  Percentage of subjects with positive SNA (≥ 100), two-fold and three-fold increasing antibodies from baseline to 28 days after the third dose

CONTACTS AND LOCATIONS:
Overall Officials: Titis Widowati, Principal Investigator — Center for Child Health Universitas Gadjah Mada (CCH-PRO UGM; Hari Wahyu N., Principal Investigator — Pediatric Research Center Universitas Sebelas Maret (PRC UNS)
Locations (21):
- Indonesia (21):
  - Dr. Moewardi District Hospital, Surakarta
  - Gajahan Primary Health Center, Surakarta
  - Gambirsari Primary Health Center, Surakarta
  - Pajang Primary Health Center, Surakarta
  - Sangkrah Primary Health Center, Surakarta
  - Sibela Primary Health Center, Surakarta
  - Bayat Primary Health Center, Yogyakarta
  - dr. Soeradji Tirtonegoro General Hospital, Yogyakarta
  - Gantiwarno Primary Health Center, Yogyakarta
  - Jogonalan 1 Primary Health Center, Yogyakarta
  - Jogonalan 2 Primary Health Center, Yogyakarta
  - Karanganom Primary Health Center, Yogyakarta
  - Kebonarum Primary Health Center, Yogyakarta
  - Kebondalem Lor Primary Health Center, Yogyakarta
  - Klaten Selatan Primary Health Center, Yogyakarta
  - Ngawen Primary Health Center, Yogyakarta
  - Pedan Primary Health Center, Yogyakarta
  - Prambanan Primary Health Center, Yogyakarta
  - Trucuk 1 Primary Health Center, Yogyakarta
  - Trucuk 2 Primary Health Center, Yogyakarta
  - Wedi Primary Health Center, Yogyakarta

IPD SHARING:
Plan to Share IPD: No